CLINICAL TRIAL: NCT03723369
Title: The Effect of Microneedling With Low Energy Laser in Androgenic Alopecia Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180301R
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Dermatologic Disease
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: accupuncture — accupuncture

SUMMARY:
Androgenetic alopecia is the most common type of hair loss in men, and affects approximately 50 percent of Caucasian men by age 50. The condition is characterized by the progressive loss of terminal hairs on the scalp in a characteristic distribution. The anterior scalp, mid scalp, temporal scalp, and vertex of the scalp are typical sites of involvement. "Male balding" and "male pattern hair loss" are additional terms used to refer to this condition.

The aim of this study is to investigate the effect of microneedling in androgenic alopecia

ELIGIBILITY:
Inclusion Criteria:

- androgenic alopecia patients

Exclusion Criteria:

* infection, immune disorder, other dermatosis in treating areas

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — androgenic alopecia
Enrollment: 7 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
hair regrowth(7-point rating scale (-3 = greatly decreased, -2 = moderately decreased, -1 = slightly decreased, 0 = no change, +1 = slightly increased, +2 = moderately increased, +3 = greatly increased).) | 12weeks
  hair regrowth(7-point rating scale (-3 = greatly decreased, -2 = moderately decreased, -1 = slightly decreased, 0 = no change, +1 = slightly increased, +2 = moderately increased, +3 = greatly increased).)

CONTACTS AND LOCATIONS:
Locations (1):
- ShinKongHospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No